CLINICAL TRIAL: NCT01337024
Title: Heart Rate Variability in Patients With Neurogenic Detrusor Overactivity Before and After Botulinum Neurotoxin Type A Intradetrusor Injections
Brief Title: Heart Rate Variability (HRV) in Patients With Neurogenic Detrusor Overactivity (NDO) Before and After Botulinum Neurotoxin Type A (BoNT/A) Intradetrusor Injections
Acronym: HRV/Botox
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Thomas M. Kessler, PD Dr. med., Neuro Urology, Spinal Cord Injury Center & Research, University of Zurich, Balgrist University Hospital
Other Study IDs: EK09/2008
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2013-01

CONDITIONS: Bladder Disorder, Neurogenic
Keywords: HRV; NDO; BoNT/A,; adverse effects
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control group: Healthy volunteers, examined with ECG without any treatment (controls)
- 100 BoNT/A: patients with neurogenic detrusor overactivity, examined with ECG, injection of 100 units BoNT/A
- 300 BoNT/A: patients with neurogenic detrusor overactivity, examined with ECG, injection of 300 units BoNT/A

SUMMARY:
Heart rate variability (HRV) is an important indicator of cardiac autonomic function and predictor of cardiac mortality and of all-cause mortality. In this study the investigators examined changes of the HRV in patients with neurogenic detrusor overactivity (NDO) undergoing botulinum neurotoxin type A intradetrusor injections (BoNT/A).

DETAILED DESCRIPTION:
BoNT/A is a common treatment in patients with NDO. Possible known side effects are urinary retention or increased post void residual. Systemic side effects seems to be rare. However this has not been investigated in detail. Although in very small amounts, BoNT/A can enter the systemic circulation during intradetrusor injections and might cause distant effects on other neuro-muscular systems, i.e. the heart. Aim of this trial is to asses potential systemic adverse effects of BoNT/A on the heart following intradetrusor injections for NDO. Potential effects on the cardiac autonomic function can be detected using HRV analysis. Patients without relevant preexisting disorders of cardiac function and proven NDO are included. During four separate visits, all subjects receive two ECG measurements before (Visit 1 and 2) and two ECG measurements following BoNT/A intradetrusor injections (Visit 3 and 4). We investigate three different groups: 1) patients not receiving BoNT/A intradetrusor injections (= control group), 2) patients receiving intradetrusor injections with 100 units BoNT/A, and 3) patients receiving intradetrusor injections with 300 units BoNT/A.

ELIGIBILITY:
Inclusion Criteria:

* patient with neurogenic detrusor overactivity
* written informed consent
* Medical indication for BoNT/A injections
* able to learn or conduct clean intermittent self-catheterization

Exclusion Criteria:

* No written informed consent
* Pregnancy
* Cancer of infection of the lower urinary tract
* Cardiac pacemaker
* Previous heart attack, angina pectoris
* Medication with effect on HRV
* Previous cardiosurgery
* Cardiac arrhythmia
* Skin disease not allowing application of ECG-electrodes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups, one control group without treatment, one group with NDO and treated with BoNT/A, both measured with ECG
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in frequency and time | The outcome measures (VLF, LF and HF, SDNN and RMSSD are measured with an ECG recording during 10 minutes, at four different time points (two times before, and two times following the BoNT/A application
  Changes in frequency (low frequency (LF), high frequency (HF), low frequency/highfrequency (LF/HF)) and time (domain parameters. This include the root mean square of differences of successive NN (normal to normal, i.e. interval between two R peaks) intervals (RMSSD), and the standard deviation of the NN intervals (SDNN)

SECONDARY OUTCOMES:
Adverse events related to BoNT/A injection (urinary tract infection, urinary retention, increasing postvoiding urine, need for intermittend catheterization | This outcome measured will be evaluated at visit 4 (six weeks, following the BoNT/A application

CONTACTS AND LOCATIONS:
Locations (1):
- Spinal Cord Injury Center & Research, University of Zürich, Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland